CLINICAL TRIAL: NCT03097289
Title: An In Vivo Recovery and Survival Study of Platelets Collected on the Trima Accel System and Stored in InterSol Solution
Brief Title: In Vivo Recovery and Survival Study of Platelets Collected on Trima Accel System and Stored in InterSol Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTS-5066
Record Dates: First submitted 2017-03-17; First posted 2017-03-31 (Actual); Results first posted 2018-11-27 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Apheresis platelets will be collected on the Trima Accel system and stored in 65% InterSol/35% plasma for all subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Platelets stored in InterSol (Experimental): Platelets collected on the Trima Accel system and stored in 65% InterSol/35% plasma
  Interventions: Device: Trima Accel system

INTERVENTIONS:
Device: Trima Accel system — A platelet apheresis procedure involves connecting the blood in the donor's vein through tubing to a machine that separates the blood components. After the separation, the desired component of the blood is removed (platelets and plasma), while the remainder of the blood components are reinfused back into the patient. To prevent clotting, an anticoagulant (ACDA) is used throughout the procedure. Following each blood collection, Platelet Additive Solution (PAS), InterSol, will be added to the platelet product to prepare the final product for 5 day storage. The entire procedure is painless and should take 90 to 120 minutes.

SUMMARY:
The purpose of this study is to evaluate the quality of platelets collected on the Trima Accel system after storage for 5 days in a Platelet Additive Solution (PAS), called InterSol.

DETAILED DESCRIPTION:
Platelets suspended in platelet additive solutions (PAS) have been collected and transfused in Europe for over 20 years. These PAS solutions outside of the United States (US) are not tied to an apheresis device; however in the US, PAS solutions have traditionally been linked to a corresponding apheresis device.

Currently in the US, there are two solutions approved by the Food and Drug Administration (FDA) as a PAS for the replacement of 65% plasma in platelet components. Isoplate Solution is approved for use with the Trima Accel® Automated Blood Collection System (Trima Accel System) and InterSol Solution is approved for use with the Amicus Separator System.

Terumo BCT is pursuing FDA clearance for InterSol in combination with the Trima Accel system in order to provide blood centers with the option to use InterSol as well as Isoplate Solution when collecting platelets to be stored in a PAS.

This is a prospective, open-label, multicenter, controlled study. Up to 40 healthy adult subjects will be enrolled in this study to ensure 24 evaluable subjects across two Investigational Sites. Evaluable is defined as the subject completing the recovery and survival procedure and neither the subject or the product meeting any of the Clinical Investigation Plan (CIP) analysis exclusion criteria.

The additional platelet donors account for screen failures, incomplete procedures and CIP exclusions.

Two (2) sets of platelets will be collected from each subject:

1. A Test unit - A hyperconcentrated platelet product collected on the Trima Accel system and diluted to a final ratio of 65% InterSol/35% plasma through the addition of InterSol directly to the platelet bag by the Trima Accel system after collection.
2. A Control sample - Fresh platelets prepared from a whole blood sample drawn from the same subject on Study Day 5 in accordance with standard procedure.

Eligible donors who have signed an informed consent will be enrolled.

SUBJECT PROCEDURES

Screening can be performed within 5 days of the apheresis procedure or combined with the Apheresis visit.

The following evaluations will be performed:

1. Informed consent will be obtained prior to initiating any study specific procedures
2. Eligibility will be confirmed
3. Demographics (age, gender, race, ethnic origin), height, and weight
4. Record medical history as per AABB criteria for healthy donors

Apheresis Visit

The following procedures will be performed:

1. Eligibility will be confirmed
2. Finger stick hemoglobin
3. Apheresis procedure

Apheresis procedures will be run according to the instructions and precautions described in the commercially available Trima Accel Operator's Manual.

The Investigator or designee will perform the venipuncture, monitor the subject during the collection, assess and provide any interventions for adverse effects, remove the needle, dress the puncture site and monitor subject through recovery.

The following information will be documented:

1. Trima procedure details
2. Adverse events (AEs)
3. Medications to treat adverse events
4. Device deficiencies

Infusion Day Visit

Five (5) days after a study subject has completed the apheresis procedure to collect Test platelets, they will return for the donation of fresh Control platelets, reinfusion of radiolabeled Test and Control platelets, and post-infusion sampling.

The following procedures will be conducted:

1. Confirm eligibility
2. Conduct pregnancy test for women of childbearing potential (serum or urine)
3. Review adverse events since the previous visit
4. Collect a whole blood sample for the production of Control platelets
5. Radiolabel Test and Control platelets and prepare for infusion
6. Infuse radiolabeled combined Test and Control platelets into subject's vein
7. Collect a 5-10 mL blood sample for pre- and post-infusion testing using the opposite arm as for the infusion

The following will be documented:

1. Vital signs (blood pressure, heart rate, temperature)
2. Adverse events
3. Medications to treat adverse events

The subject will return to the study site daily (except on weekends) between Study Day 6 and Study Day 12 . A total of 5 blood samples are required to be collected in this 7 day period in order for the subject's data to be evaluable. The subject will also return to the study site for a final visit on Study Day 16.

At each of these visits a blood sample will be collected for testing.

The following will be documented:

1. Adverse events
2. Medications to treat adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Normal health status as per AABB criteria for a healthy donor
3. Able to commit to the study schedule
4. Meets the inclusion criteria defined by the Blood Center for an apheresis platelet with PAS collection on the Trima Accel system. These criteria are based on FDA Regulations and AABB standards. Note: Participants who are deferred from volunteer community donations because of travel restrictions, piercings, or tattoos may participate in the study, as products are not transfused
5. Participants of child-bearing potential (either male or female) must agree to use an effective method of contraception during the course of the study
6. Female of childbearing potential must be willing to take a pregnancy test prior to infusion of radiolabeled platelets
7. Has given written informed consent

Exclusion Criteria:

1. Previously received radiation therapy
2. Has been diagnosed with a platelet disorder (ie, platelet dysfunction)
3. Already participated in 4 research studies involving radioisotopes within the contemporaneous calendar-year
4. Pregnant or nursing females
5. Participation currently, or within the last 12 months, in another investigational trial that would potentially interfere with the analysis of this investigation
6. History of known hypersensitivity to indium or chromium
7. Treatment with aspirin or aspirin containing medications within 7 days of apheresis or treatment with non-steroidal anti inflammatory drugs (NSAID), anti-platelet agents or other drugs affecting platelet viability within 3 days of apheresis (eg, ibuprofen or other NSAIDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cancelas, MD, PhD, Principal Investigator — Hoxworth Blood Center; Mehraboon S Irani, MD, Principal Investigator — Versiti Blood Health
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - BloodCenter of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A participant was considered "enrolled" upon signing the informed consent form.
Pre-assignment Details: 33 participants consented/enrolled: 1 screen-failed; 32 participants started an apheresis procedure and were therefore included in the Safety Analysis Set
  6 participants did not complete all study procedures, resulting in 26 participants completing the study; 2 participants met the Full Analysis set exclusion criteria
  24 = Full Analysis set
Groups:
- Platelets Stored in InterSol: Healthy adult volunteer blood donors will undergo apheresis for a single hyperconcentrated platelet product. Platelets will be stored in 65% InterSol/35% plasma for 5 days. Following storage for 5 days, an aliquot of Test platelets will be radiolabeled with either 111In or 51Cr. Similarly an aliquot of freshly prepared platelets derived from a whole blood sample donated on Day 5 (Control) will be tagged with the radiolabel not used in the Test platelets. The labeled aliquots will then be infused simultaneously on Day 5 back to the autologous donor.
Period: Overall Study
Arm/Group | Platelets Stored in InterSol
Started | 32
Completed | 26
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Equipment failure | 2
Not completed — Collected platelet product unusable | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set = Includes all participants who underwent any study related apheresis procedure, defined as having had venipuncture for apheresis.
Arm/Group | Platelets Stored in InterSol
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  Age ≥ 18 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 31
Region of Enrollment [Number; unit: participants]
  United States | 32
Height [Mean (Standard Deviation); unit: inches] | 68.3 (3.24)
Weight [Mean (Standard Deviation); unit: pounds] | 196.5 (48.27)

OUTCOME MEASURES:

1. Primary Outcome: Recovered Percentage of the Extrapolated Platelet Count at Time 0
Description: The percent recovery of platelets stored in InterSol for 5 Days as compared to fresh controls. Percent recovery was expressed as a percentage and was extrapolated for a value at Time 0. The FDA acceptance criteria for recovery is >66% of control with a 1-sided 97.5% confidence limit.
Time Frame: 11 days (+/- 1 day)
Population: The Full Analysis Set (FAS) consisted of all completed procedures/products where the corresponding Test and Control values for primary endpoint were valid. Data points could be excluded from FAS if:
  1. Primary endpoint laboratory samples were lost/not available
  2. Failure of site to follow post-collection handling procedures for endpoint assays
Measure: Mean (Standard Deviation); unit: percent of extrapolated platelet count
Groups:
- Test Platelets Collected and Stored in InterSol: Platelets stored in InterSol
  One Test unit will be collected as a hyperconcentrated platelet product. The Test unit will be diluted to a final ratio of 65% InterSol/35% plasma and stored for 5 days.
- Control Platelets: Control Platelets
  An aliquot of freshly prepared platelets derived from a whole blood sample.
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets
Number analyzed (Participants) | 24 | 24
percent of extrapolated platelet count | 45.15 (12.256) | 56.02 (13.162)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets; Test type: Non-Inferiority — The acceptance criterion for the recovery (%) of platelets is the demonstration of non-inferiority by the rejection of the Null Hypothesis (H0) defined by the following hypotheses: Null Hypothesis H0: μd ≤ 0 where μd=μT-0.66*μC Alternate Hypothesis H1: μd > Let Xi = (XTi-0.66*XCi) be a difference if recovery for patient i. The sample mean and standard deviations of these observed differences will be used to construct the lower limit of a 1-sided 97.5% confidence interval; Mean Difference (Final Values) = 8.18, 97.5% CI 1-sided [lower limit 4.03]

2. Primary Outcome: Number of Days of Platelet Survival
Description: Survival of platelets stored in InterSol for 5 Days as compared to fresh controls. Survival was expressed in days and was approximated using linear regression. The FDA acceptance criteria for survival is >58% of control with a 1-sided 97.5% confidence limit
Time Frame: 11 days (+/- 1 day)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Test Platelets Collected and Stored in InterSol | Control Platelets
Number analyzed (Participants) | 24 | 24
days | 5.40 (0.991) | 7.93 (1.483)
Statistical Analysis 1: Comparison: Test Platelets Collected and Stored in InterSol vs Control Platelets; Test type: Non-Inferiority — The acceptance criterion for the survival (days) of platelets is the demonstration of non inferiority by the rejection of the null hypothesis (H0) defined by the following hypotheses: Null Hypothesis H0: μd ≤ 0 where μd = μT-0.58 × μC Alternate Hypothesis H1: μd > 0; Mean Difference (Final Values) = 0.80, 97.5% CI 1-sided [lower limit 0.39]

ADVERSE EVENTS:
Time Frame: Adverse events that occurred on or after the start of the apheresis procedure (time of venipuncture) until study completion (16 days +/- 1 day).
Description: Treatment emergent adverse events were analyzed in the Safety Analysis set. Treatment began with the apheresis venipuncture.
Arm/Group | Platelets Stored in InterSol
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 6/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Platelets Stored in InterSol (N=32)
Injection site extravasation (General disorders) | 4
Paraesthesia oral (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retains the right to review and comment on any public disclosure of study results. If no response is received within 60 days, the Principal Investigator may presume that the submission for publication may proceed without delay. If the Sponsor asks to defer publication, Study Site shall not publish, or otherwise disclose to any third party, any of the information contained in the publication or presentation until expiration of the 60 day period.

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03097289/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03097289/SAP_001.pdf